CLINICAL TRIAL: NCT06373692
Title: REspiratory diSEAse cohoRt Studies of CHinese Medicine for Asthma (RESEARCH- Asthma)
Status: Not yet recruiting | Type: Observational
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Collaborators: The First Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other); Tianjin University of Traditional Chinese Medicine (Other); Third Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other); Hebei Provincial Hospital of Traditional Chinese Medicine (Other Government); Peking University People's Hospital (Other); The Affiliated Hospital of Jiangxi University of Traditional Chinese Medicine (Other); The First Affiliated Hospital of Zhengzhou University (Other); Affiliated Hospital of Liaoning University of Traditional Chinese Medicine (Other); The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: TCM for Asthma Cohort
Record Dates: First submitted 2024-01-03; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Bronchial Asthma
Keywords: Bronchial asthma; Asthma control rate; Number of acute attacks; Cohort studies
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The biological samples include serum samples, plasma samples, urine samples, sputum samples, and exhaled air condensate samples.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Traditional Chinese Medical cohort: The standardized use of TCM treatment regimen was regarded as an exposure factor, and the treatment methods of the enrolled patients were defined and grouped: patients who took medication continuously for more than 3 months per year, or who took medication intermittently for more than 6 months in the total time of the year, were in the exposure group.
- Non Traditional Chinese Medical cohort: Those who used conventional Western medicine treatment without using standardized Chinese medicine treatment regimen were in the non-exposure group.

SUMMARY:
The purpose of this study is to define the standard use of TCM treatment regimen as the TCM cohort group and the non-TCM cohort group of those who use conventional Western medicine treatment without the standard TCM treatment regimen through a multi-center, large-sample prospective cohort study design. To evaluate the clinical efficacy and safety of TCM treatment regimens in the treatment of bronchial asthma, and to provide high-quality evidence for the promotion and application of TCM syndrome differentiation treatment in bronchial asthma.

DETAILED DESCRIPTION:
Bronchial asthma is characterized by chronic inflammation of the airways, which is often recurrent, long-lasting and difficult to cure. Clinical studies have confirmed that the clinical symptoms and quality of life of asthma patients have been significantly improved after TCM intervention. However, most of the current clinical research methods on asthma are small-sample and RCT studies, resulting in insufficient demonstration of efficacy, and there is an urgent need to carry out multi-center, large-sample, high-quality real-world studies in order to obtain higher quality evidence-based medical evidence.

This is a multi-center, large-sample prospective cohort study, which will evaluate the clinical efficacy and safety of TCM treatment regimens in the treatment of bronchial asthma, and provide high-quality evidence for the promotion and application of TCM syndrome differentiation therapy in bronchial asthma. The cohort study will enroll 1508 patients, and the standard use of TCM treatment regimen will be set as the TCM cohort group, and those who will use the conventional treatment of Western medicine but not the standard TCM treatment regimen will be the non-TCM cohort group. The asthma control rate was the main outcome index, and the asthma control questionnaire (ACQ), asthma quality of life score (AQLQ), clinical symptom and sign score, lung function, exhaled nitric oxide, induced sputum inflammation phenotype, glucocorticoid dose, and fast-acting β2 agonist dose were the secondary outcome indicators. Follow-up was conducted every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the diagnosis of bronchial asthma;
2. Age 18~80 years old;
3. Have not participated in other clinical studies within 1 month before enrollment;
4. Voluntarily participate in the study and sign the informed consent form.

Exclusion Criteria:

1. Patients with respiratory failure and mechanical ventilation during acute asthma exacerbation;
2. Delirium, impaired consciousness, dementia, and various mental illnesses;
3. Patients with other lung diseases such as COPD, lung abscess, cystic fibrosis, bronchiectasis, etc., and severe liver and kidney diseases;
4. Patients with neuromuscular diseases that affect respiratory motor function and are unable to complete the six-minute walk test;
5. Pregnant and lactating patients;
6. Those who are participating in other clinical trials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are eligible for a diagnosis of bronchial asthma disease
Sampling Method: Non-Probability Sample
Enrollment: 1508 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Asthma control rate | The follow-up period was followed up every 3 months for 1 year.
  According to the composite indicators such as symptoms, medication and pulmonary function test results, the clinical control level of asthma was divided into complete control, partial control and uncontrolled, and the asthma control rate of patients was evaluated according to the clinical control level of asthma.

SECONDARY OUTCOMES:
Number of exacerbations | The follow-up period was followed up every 3 months for 1 year.
  The number of acute attacks is mainly recorded
Asthma exacerbation severity | The follow-up period was followed up every 3 months for 1 year.
  Worsening lung function during asthma attacks is characterized by decreased expiratory flow, and the severity of the exacerbation can be graded by the patient's symptoms, lung function, and arterial blood gas analysis.According to the frequency of daytime and nighttime asthma attacks and pulmonary function test results, the patients were divided into 4 grades, namely: 1 intermittent attack; 2 mild persistent; 3 moderate persistent and 4 severe persistent.The severity of the asthma attack was assessed using a rating scale.
Change in severity of chronic persistent disease | The follow-up period was followed up every 3 months for 1 year.
  Although the patient does not have an acute attack of asthma, there are still symptoms such as wheezing, cough, chest tightness and other symptoms with different frequency and degrees for a long time, which may be accompanied by decreased pulmonary ventilation function. The severity of chronic persistent asthma can be classified into four levels: intermittent, mildly persistent, moderately persistent, and severely persistent, according to the frequency of daytime and nighttime asthma symptoms and the results of pulmonary function tests.The severity of the asthma attack was assessed using a rating scale.
The dose used by glucocorticoids | The follow-up period was followed up every 3 months for 1 year.
  Corticosteroids are the drug of choice for long-term asthma treatment. The vast majority of patients with chronic persistent asthma are well controlled by inhaling low-dose corticosteroids (equivalent to 400 micrograms of budesonide per day).
Rapid-acting beta2 agonists use drugs and doses | The follow-up period was followed up every 3 months for 1 year.
  Beta2 agonists are asthma drugs that stimulate beta2 receptors distributed on airway smooth muscle to produce bronchodilating effects. These drugs are bronchodilators and are the drugs of choice for acute asthma attacks (airway spasm), which can quickly improve symptoms such as dyspnea, cough, etc. If given by inhalation, salbutamol 100-200mcg or terbutaline 250-500mcg at a time and repeat every 20 minutes if necessary.
Asthma Control Test (ACT) score | The follow-up period was followed up every 3 months for 1 year.
  The ACT score correlates well with the level of asthma control in patients as assessed by experts. The questionnaire included wheezing symptoms, activity limitations, frequency of use of rescue medication, patients' asthma control and self-assessment, with a total of 5 items. Each item is scored on a scale of 1~5, with a total score of 5~25 points, and the higher the score, the better the control of asthma symptoms.
Asthma Control Questionnaire (ACQ) | The follow-up period was followed up every 3 months for 1 year.
  The ACQ questionnaire will measure the quality of life associated with asthma. The ACQ questionnaire consists of either 7 questions (ACQ-7) or 6 questions (ACQ-6). In questions 1-6, patients recalled their experiences from the previous 7 days and answered using a scale of 7 (from 0 = complete control to 6 = very poor control). The seventh question refers to % FEV1 of the reference value and must be completed by the staff of the website. The questionnaire score is the average of either 7 responses (ACQ-7) or 6 responses (ACQ-6). The score is interpreted as follows: 0.75 or less: adequate asthma control. From 0.75 to 1.50: partially controlled asthma. Over 1.50: inadequate asthma control.
Asthma Quality of Life Score (AQLQ) | The follow-up period was followed up every 3 months for 1 year.
  It is used to measure the severity of asthma and its impact on patients' quality of life, including 35 items in 5 aspects. The AQLQ score relates to activity limitation, asthma symptoms, psychological condition, response to stimuli, and concern for one's own health, and the form assesses the degree of impact of asthma on a 7-point scale, with a maximum impact of 1 point and no impact of 7 points.
Anxiety Self-Assessment Form (SAS) | The follow-up period was followed up every 3 months for 1 year.
  It included 20 items reflecting the subjective feelings of anxiety, and each item was divided into four levels according to the frequency of symptoms, including 15 positive scores and 5 reverse scores. The cut-off value for the standard deviation of SAS is 50 points, with higher scores indicating more severe symptoms of anxiety.Among them, 50 to 59 are classified as mild anxiety, 60 to 69 are classified as moderate anxiety, and more than 69 are severe anxiety.
Depression Self-Rating Scale (SDS) | The follow-up period was followed up every 3 months for 1 year.
  The SDS Depression and Anxiety Test Form contains 20 items, which are scored on a 4-point scale, with 1 indicating occasional symptoms, 2 indicating sometimes symptoms, 3 indicating frequent symptoms, and 4 indicating persistent symptoms. A rough score is obtained by adding the scores in each of the 20 items. Multiply the rough score by 1.25 and then take the integer part to get the standard score. Generally speaking, depression with a total score of less than 52 is normal, 53-62 is mild depression, 63-72 is moderate depression, and 72 or more is severe depression. The higher the score, the more severe the symptoms.
Pulmonary function | The follow-up period was followed up every 3 months for 1 year.
  FVC, FEV1, FEV1 % of the estimated value, FEV1/FVC were mainly used for evaluation.
Exhaled nitric oxide (FeNO) | The follow-up period was followed up every 3 months for 1 year.
  The measuring instrument uses an exhaled nitric oxide measurement system to record the FeNO value of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Jian-sheng Li, Professor, Study Chair — The First Affiliated Hospital of Henan University of Traditional Chinese Medicine
Locations (1):
- The First Affiliated Hospital of Henan University of Traditional Chinese Medicine, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No